CLINICAL TRIAL: NCT05963425
Title: The Effects on Physical Activity on Mitochondrial Function in Skin Fibroblasts in Patients with Parkinson's Disease: a Study Protocol.
Brief Title: The Effects on Physical Activity on Mitochondrial Function in Skin Fibroblasts in Patients with Parkinson's Disease.
Acronym: PARKEX
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ramon Llull (Other)
Collaborators: University of Coimbra (Other); Hospital Vall d'Hebron (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PARKEX
Record Dates: First submitted 2023-07-12; First posted 2023-07-27 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-01

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Physical Activity; Mitochondrial Function; Skin Fibroblasts
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Physical activity: basic physical training (BPT) (Experimental): Exercises will target the large muscle groups, with a component/emphasis on the eccentric phase of concentration. The kBox4 Platform (Exxentric AB), a device designed to maximize performance and training outcomes, will be used to enhance the eccentric phase of the exercises.
  kBox4 is controlled by a specific program, Kmeter, which records and stores all the information (duration, intensity, repetitions, etc.) of each movement. Exxentric kBox4 will be adapted with special harnesses, insurances on the wall and in front of support bars, according to the needs of the patients. In addition to the major muscle groups, specific attention will be given to the key muscles involved in the gait cycle, such as the tibialis anterior, medial gastrocnemius, rectus femoris, and hamstrings, from a biomechanical perspective.
  Interventions: Other: Physical activity
- Physical activity: BPT combined with functional exercises (Experimental): In addition to the BPT program (which includes the transverse focus on strength and resistance exercises), this intervention group will incorporate functional exercises that involve dual task training. The dual task training can encompass both motor-motor and motor-cognitive activities. This means that coordinated exercises will be performed, with cognitive activities introduced at the extremes of the movement. This approach ensures engagement of both physical and cognitive abilities during the PA sessions.
  Interventions: Other: Physical activity
- Control (Active Comparator): Participants in the control group will maintain their regular daily routines throughout the study period.
  Interventions: Other: usual clinical practice

INTERVENTIONS:
Other: Physical activity — This physical activity program will be based only on the work of basic physical training, in which specifically and mainly the strength and resistance will be worked, but also flexibility
  Other Names: Exercise
  Arms: Physical activity: BPT combined with functional exercises; Physical activity: basic physical training (BPT)
Other: usual clinical practice — usual clinical practice
  Arms: Control

SUMMARY:
The aim of this study is to investigate the effect of physical activity on mitochondrial function in skin fibroblasts in patients with Parkinson's disease.

DETAILED DESCRIPTION:
A randomized double-blind clinical trial will be conducted to study the effects of physical activity on mitochondrial function in skin fibroblasts in patients with Parkinson's disease. It is an intervention study, and twenty-four patients will be needed. Once the subjects have been selected, they will be randomly assigned into three groups (eight patients in each group). The first group will perform basic physical training (BPT) based on strength and resistance, the second group will perform BPT combined with functional exercises (BPTFE) with cognitive and motor training, and the third group will not carry out any activity program, serving as control. The interventions will last 60 minutes, with a frequency of 3 times a week, during 16 weeks. The control group will receive 4 months of PA from the program that has obtained the best results,in terms of symptoms and quality of life, after the last evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a medical diagnosis of idiopathic PD, Hoehn and Yahr scale stages of I-III.
* Patients who score ≥26 on the Montreal Cognitive Assessment (MoCA).
* Patients who have signed the IC.
* Patients with stable medication.
* Age between 50 and 70 years, and able to walk independently for 6 minutes.

Exclusion Criteria:

* Patients with a pathology other than idiopathic PD.
* Patients with cognitive impairment (MoCA <26 points).
* Patients with uncontrolled cardiovascular disease, visual impairment, or recent musculoskeletal disorders in the extremities.
* Patients who are performing another therapeutic exercise protocol.
* Patients who have undergone surgery to influence any symptom from the PD.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in oxygen consumption rate | Beginning of the study and after 4 months
  Oxygen uptake (VO2, mlkg-1min-1) measured by Seahorse XFe96
Change in ATPmax levels | Beginning of the study and after 4 months
  Maximal mitochondrial ATP production rates measured by Seahorse XFe96

SECONDARY OUTCOMES:
Non-motor and motor function | Beginning of the study, first visit
  non-motor and motor experiences of daily living and motor complications measured by the MDS-Sponsored Revision of the UPDRS (MDS-UPDRS) questionnaire
Sleepiness | Beginning of the study, first visit
  Self-administered questionnaire with 8 questions measured by the Epworth Sleepiness Scale (ESS) questionnaire
Mobility | Beginning of the study, first visit
  clinical performance-based measure of lower extremity function, mobility and fall risk, measured by the Timed Up and Go Test (TUG) questionnaire
Cognitive aspects | Beginning of the study, first visit
  Cognitive aspects measured by the Montreal Cognitive Assessment scale (MoCA)
Mood | Beginning of the study, first visit
  Intensity of depression in clinical and normal patients measured by the Beck Depression Inventory (BDI) questionnaire
Non-motor and motor function | End of the study (4 Months)
  non-motor and motor experiences of daily living and motor complications measured by the MDS-Sponsored Revision of the UPDRS (MDS-UPDRS) questionnaire
Sleepiness | End of the study (4 Months)
  Self-administered questionnaire with 8 questions measured by the Epworth Sleepiness Scale (ESS) questionnaire
Mobility | End of the study (4 Months)
  clinical performance-based measure of lower extremity function, mobility and fall risk, measured by the Timed Up and Go Test (TUG) questionnaire
Cognitive aspects | End of the study (4 Months)
  Cognitive aspects measured by the Montreal Cognitive Assessment scale (MoCA)
Mood | End of the study (4 Months)
  Intensity of depression in clinical and normal patients measured by the Beck Depression Inventory (BDI) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Joel Montane, PhD, Principal Investigator — Universitat Ramon Llull
Locations (1):
- Vall Hebron Institut de Recerca, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Magana JC, Deus CM, Gine-Garriga M, Montane J, Pereira SP. Exercise-Boosted Mitochondrial Remodeling in Parkinson's Disease. Biomedicines. 2022 Dec 12;10(12):3228. doi: 10.3390/biomedicines10123228. PMID 36551984
- [Background] Deus CM, Pereira SP, Cunha-Oliveira T, Pereira FB, Raimundo N, Oliveira PJ. Mitochondrial remodeling in human skin fibroblasts from sporadic male Parkinson's disease patients uncovers metabolic and mitochondrial bioenergetic defects. Biochim Biophys Acta Mol Basis Dis. 2020 Mar 1;1866(3):165615. doi: 10.1016/j.bbadis.2019.165615. Epub 2019 Nov 20. PMID 31759069
- [Derived] Magana JC, Deus CM, Baldellou L, Avellanet M, Gea-Rodriguez E, Enriquez-Calzada S, Laguna A, Martinez-Vicente M, Hernandez-Vara J, Gine-Garriga M, Pereira SP, Montane J. Investigating the impact of physical activity on mitochondrial function in Parkinson's disease (PARKEX): Study protocol for A randomized controlled clinical trial. PLoS One. 2023 Nov 22;18(11):e0293774. doi: 10.1371/journal.pone.0293774. eCollection 2023. PMID 37992028